CLINICAL TRIAL: NCT03729050
Title: Rehabilitation Coordinators in Specialist Psychiatry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Ingrid Anderzen, Associate professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REKO-A
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Mental Disorder; Rehabilitation
Keywords: Mental Disorder; Rehabilitation
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention with rehabilitation coordinator (Experimental)
  Interventions: Behavioral: Rehabilitation Coordinator in Specialist Psychiatry
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Rehabilitation Coordinator in Specialist Psychiatry — Rehabilitation Coordinator service in Specialist Psychiatry
  Arms: Intervention with rehabilitation coordinator

SUMMARY:
REKO-A is a randomized controlled intervention study that addressed women and men on sick leave in Uppsala County. Participants which are on sick leave due to mental illness.

ELIGIBILITY:
Inclusion Criteria:

* Be on sick leave
* Have moderate to severe affective and / or moderate / severe anxiety disorder, such as: Bipolar disorder, depression, posttraumatic stress disorder, generalized anxiety disorder, neuropsychiatric disability
* Enrolled at the Academic hospital in Uppsala

Exclusion Criteria:

* High suicidal risk
* Extensive somatic disorders (somatic multichannel)
* Patients outside Uppsala County
* Taking part in an ongoing vocational rehabilitation

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-10-24 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Return to work (RTW)/entry into work or studies | 1 year
  Number of Participants that have RTW/entry into work or studies
Magnitude of sick leave | 1 year
  Proportion of sick leave in the study population
Length of sick leave | 1 year
  Sick leave duration

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala university, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersen A, Berglund E, Anderzen I. Rehabilitation coordinator intervention versus control in psychiatric specialist care for return to work and reduced sick leave: study protocol of a randomised controlled trial. BMC Public Health. 2020 Feb 19;20(1):250. doi: 10.1186/s12889-020-8238-3. PMID 32075611